CLINICAL TRIAL: NCT06364189
Title: Unraveling the Mechanisms of a Novel Music Intervention for Physical Activity Promotion in Older Adults
Brief Title: Inspiring Seniors Toward Exercise Promotion
Acronym: iSTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Greensboro (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jennifer L. Etnier, Distinguished Professor, University of North Carolina, Greensboro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FY22-119; R61AG084479 (NIH)
Record Dates: First submitted 2024-03-29; First posted 2024-04-15 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Cognitively Normal Older Adults
Keywords: music; aerobic exercise; strength training; cognitive performance
MeSH Terms: interventions — Music Therapy; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and music stimulation (Experimental): Participants are given an aerobic and strength training program with faded supervision across 6 months.
  For aerobic exercise (AE), participants will be instructed to walk at moderate intensity with duration increasing up to an ultimate goal of 150 min/week. Participants will be trained to walk in synchrony with the beats of their personalized playlists.
  The strength training (ST) incorporates single-leg exercises for balance training and training with resistance bands and body weight. During the ST, participants will be asked to synchronize their concentric and eccentric muscle contractions in time with the tempo of BMS playlists at a specific beats-per-minute rhythm.
  Interventions: Behavioral: Music; Behavioral: Exercise
- Exercise only (Active Comparator): Participants are given an aerobic and strength training program with faded supervision across 6 months.
  The ST incorporates single-leg exercises for balance training and training with resistance bands and body weight.
  For aerobic exercise (AE), participants will be instructed to walk at moderate intensity with duration increasing up to an ultimate goal of 150 min/week.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Music — Individualized play lists of music with the beats accentuated will be developed at a range of cadences. The music intervention is such that during strength training participants will be asked to sync their concentric and eccentric muscle contractions in time with the tempo of playlists. For aerobic exercise (AE), the tempo of playlists will be adjusted to match individual walking cadence for participants to be trained to walk in sync with the beats of the playlists.
  Arms: Exercise and music stimulation
Behavioral: Exercise — The ST incorporates single-leg exercises for balance training and training with resistance bands and body weight.
  For aerobic exercise (AE), participants will be instructed to walk at moderate intensity with duration increasing up to an ultimate goal of 150 min/week.

SUMMARY:
The goal of this clinical trial is to test the benefits of beat-accented music stimulation (BMS) for behavioral changes of physical activity (PA) in older adults. Specific Aims are to determine (1) whether BMS beneficially influences PA behaviors and psychological responses to PA in older adults for 6 months, and (2) whether exercising with BMS differently influences physical and cognitive functioning as well as quality of life in older adults.

To test the effects of BMS on PA, participants will be randomly assigned to an exercise intervention that either includes BMS or does not include BMS. Participants will attend a supervised group strength training (ST) (30 min/day) and aerobic exercise (AE) (30-50 min/day) session for 3 days/week for the first 2 months, 1 day/week for the next 2 months (while encouraging participants to independently perform both AE and ST on other days), and independently for the final 2 months (always with a goal of performing >150min/week AE and 3 days/week of ST for 30 min/day.

ELIGIBILITY:
Inclusion Criteria:

* At least 65 years old.
* Ambulatory/capable of walking for 6 minutes without pain or aid such as a walker/cane.
* Able to speak and read English.
* Healthy enough to exercise at moderate intensity with or without medical clearance by a primary care physician.
* Living in the community for the duration of the study (6 months).
* Having a reliable means of transportation.
* Having a safe place (at least 6 feet by 6 feet of open space) at home for unsupervised exercise training.
* Having no diagnosis or symptoms of cognitive impairment.
* Having no symptoms of suicidal ideation and not meeting criteria for depressive disorder.
* Physically low-active by doing < 60 min/week of moderate-intensity aerobic exercise and no strength training for the last 3 months.

Exclusion Criteria:

* Diagnosis of neurological disorder or spinal cord disorder.
* Known exercise contraindications.
* Current cancer treatment.
* Stroke or neural impairment in the past 6 months.
* Hip/knee/spinal fracture or surgery in the past 6 month.
* Unable or unwilling to attend intervention classes 3x/week in Months 1-2 and 1x/week in Months 3-4.
* Currently participating in any other physical activity or fitness-related research study.
* Use of medication for Alzheimer's disease.
* Change in dosage of medications prescribed for anxiety or depression within the previous 6 months.
* Regularly drink > 14 alcoholic beverages a week or current illicit drug use.
* Having no diagnosis or symptoms of cognitive impairment.
* Meet the threshold for clinical depression.
* Uncorrected hearing or visual impairments.
* Unable to understand the study procedures.
* One of the household members is participating in this study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Physical activity (objective) | Accelerometers will be worn for 4 days at baseline and months 1, 2, 3, 4, 5, and 6.
  Physical activity behavior assessed using accelerometry
Ecological Momentary Assessment (EMA): Affective response to PA | Will be collected using EMA for 4 days at baseline and months 1, 2, 3, 4, 5, and 6.
  Captures the shift in core affective valence (feeling good vs bad) from pre-PA to during-PA.
Ecological Momentary Assessment (EMA): Perceived autonomy | Will be collected using EMA for 4 days at baseline and months 1, 2, 3, 4, 5, and 6.
  Assesses participant's perceived autonomy over exercise behavior.
Ecological Momentary Assessment (EMA): Perceived exertion | Will be collected using EMA for 4 days at baseline and months 1, 2, 3, 4, 5, and 6.
  Assesses participant's perceived exertion during PA.
Ecological Momentary Assessment (EMA): Behavioral intention | Will be collected using EMA for 4 days at baseline and months 1, 2, 3, 4, 5, and 6.
  Assesses degree to which participant intends to engage in PA.
Ecological Momentary Assessment (EMA): Physical Activity setting | Will be collected using EMA for 4 days at baseline and months 1, 2, 3, 4, 5, and 6.
  Assessed the physical and social setting in which a participant engages in physical activity.
Ecological Momentary Assessment (EMA): Anticipated, remembered, and incidental affect | Will be collected using EMA for 4 days at baseline and months 1, 2, 3, 4, 5, and 6.
  Will assess how participant expects to feel after engaging in PA, how participant remembers feeling after engaging in PA, and how participant currently feels.
Ecological Momentary Assessment (EMA): Social Support for Exercise | Will be collected using EMA for 4 days at baseline and months 1, 2, 3, 4, 5, and 6.
  Measures with whom a person is exercising
Physical activity (self-report) | Will be reported daily from the first day of the intervention to the last day of the intervention (6 months)
  Aerobic exercise and strength training self-reported

SECONDARY OUTCOMES:
Cognitive performance - General | At pre-test and following study completion (approximately 6 months after pre-test)
  Assessed using the Montreal Cognitive Assessment. Scores range from 0-30 with a higher score indicative of a better outcome.
Cognitive performance - Tower of London | At pre-test and following study completion (approximately 6 months after pre-test)
  Assessed using the Tower of London test. Both accuracy and reaction time are recorded with higher scores for accuracy and lower scores for reaction time indicative of a better outcome.
Cognitive performance - NIH Toolbox Oral Reading Recognition Test | At pre-test and following study completion (approximately 6 months after pre-test)
  Assessed using the NIH Toolbox Oral Reading Recognition Test
Cognitive performance - NIH Toolbox List Sort Working Memory Test | At pre-test and following study completion (approximately 6 months after pre-test)
  Assessed using the NIH Toolbox List Sort Working Memory Test
Cognitive performance - NIH Toolbox Picture Sequence Test | At pre-test and following study completion (approximately 6 months after pre-test)
  Assessed using the NIH Toolbox Picture Sequence Test
Cognitive performance - NIH Toolbox Dimensional Change Card Sort Test | At pre-test and following study completion (approximately 6 months after pre-test)
  Assessed using the NIH Toolbox Dimensional Change Card Sort Test
Cognitive performance - NIH Toolbox Flanker Inhibitory Control and Attention Test | At pre-test and following study completion (approximately 6 months after pre-test)
  Assessed using the NIH Toolbox Flanker Inhibitory Control and Attention Test
Cognitive performance - Mnemonic Similarity Task | At pre-test and following study completion (approximately 6 months after pre-test)
  Assessed using the Mnemonic Similarities Task
Cognitive performance - Perceptual Discrimination Task | At pre-test and following study completion (approximately 6 months after pre-test)
  Assessed using the Perceptual Discrimination Task
Health Related Quality of Life | At pre-test and following study completion (approximately 6 months after pre-test)
  Assessed using the RAND 36-Item Short-Form Health Survey with scores ranging from 0-100 and a higher score being indicative of a better outcome.
Physical activity (subjective) | At pre-test and following study completion (approximately 6 months after pre-test)
  Physical activity behavior is assessed using the Physical Activity and Sedentary Behavior Questionnaire (PASB-Q) which includes open-ended questions to assess frequency of physical activity and multiple choice questions to assess perceived fitness and sedentary behaviors.
Music Reward Experience | At pre-test and following study completion (approximately 6 months after pre-test)
  Music Reward Experience will be assessed using the Barcelona Music Reward Questionnaire (BMRQ) which uses a 5-point Likert scale. Responses are converted to z-scores which are then combined into factor scores and converted into T-scores ranging from 0-100 with a higher score meaning a more positive experience.
Treatment Satisfaction | At pre-test and following study completion (approximately 6 months after pre-test)
  Treatment Satisfaction will be assessed using the Client Satisfaction Questionnaire (CSQ-8) with scores ranging from 8-32 and a higher score being indicative of a better outcome.
Body Mass Index | At pre-test and following study completion (approximately 6 months after pre-test)
  Body mass index will be assessed as a ratio of weight to height with measurements taken in the lab setting.
Waist/Hip/Leg Circumference | At pre-test and following study completion (approximately 6 months after pre-test)
  Waist/Hip/Leg Circumference will be assessed using a measuring tape.
Sagittal Diameter | At pre-test and following study completion (approximately 6 months after pre-test)
  Sagittal Diameter will be assessed using a measuring tape.
Blood Pressure | At pre-test and following study completion (approximately 6 months after pre-test)
  Systolic and diastolic blood pressure will be assessed using an automated blood pressure cuff.
Handgrip Strength | At pre-test and following study completion (approximately 6 months after pre-test)
  Handgrip Strength will be assessed using a goniometer.
Timed Up and Go (TUG) | At pre-test and following study completion (approximately 6 months after pre-test)
  Timed Up and Go (TUG) will be assessed using standard instructions asking participants to stand up from a seated position, to walk 3-meters, turn around, return 3-meters, turn around, and sit back down. Performance is the time needed to complete the task.
10-Meter Walk | At pre-test and following study completion (approximately 6 months after pre-test)
  10-Meter Walk will be assessed with a stop watch over a clearly marked 10-meter distance.
4-Stage Balance Test | At pre-test and following study completion (approximately 6 months after pre-test)
  4-Stage Balance Test will be assessed using standard directions. Duration of the ability to stand in 4 different poses with eyes open and without changing posture.
6-Minute Walk Test (6MWT) | At pre-test and following study completion (approximately 6 months after pre-test)
  6-Minute Walk Test (6MWT) will be assessed as the distance travelled in 6-minutes around a clearly marked space in a gymnasium.
30-second Chair Stand | At pre-test and following study completion (approximately 6 months after pre-test)
  The number of sit-to-stand maneuvers that can be completed within 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Etnier, PhD, Principal Investigator — University of North Carolina, Greensboro; Kyoungshin Park, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - University of North Carolina at Greensboro, Greensboro, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park KS, Williams DM, Etnier JL. Exploring the use of music to promote physical activity: From the viewpoint of psychological hedonism. Front Psychol. 2023 Jan 25;14:1021825. doi: 10.3389/fpsyg.2023.1021825. eCollection 2023. PMID 36760458